CLINICAL TRIAL: NCT04694443
Title: Feasibility and Cost-effectiveness of a Multidisciplinary Home-based Telehealth Intervention Program to Reduce Falls in Parkinson´s Disease (TeleFall).
Brief Title: Multidisciplinary Home-based Tele-rehabilitation Intervention
Acronym: TeleFall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esther Cubo (Other)
Collaborators: Hospital Universitario de Burgos (Other); Instituto de Salud Carlos III (Other Government); University of Burgos (Unknown)
Responsible Party: Sponsor-Investigator, Esther Cubo, MD, PhD, Principal Investigator, Hospital Universitario de Burgos
Organization: Hospital Universitario de Burgos (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI19/00670
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
Keywords: Falls; Cost-effectiveness; Qaly
MeSH Terms: conditions — Parkinson Disease | interventions — Physical Therapy Modalities; Neurologists; Nurses; Educational Status

STUDY DESIGN:
Intervention Model Description: Single blind, randomized, case-control study
Who Masked: Outcomes Assessor
Masking Description: The rater will be blind to the patient status (study vs. control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): The study group will receive the multidisciplinary tele-health intervention plus standard medical care
  Interventions: Procedure: Multidisciplinary tele-health intervention (physical therapy, neurologist, nurse, psychologist)
- Control group (Placebo Comparator): The control group will receive the best standard medical care
  Interventions: Other: Standard in-office medical care

INTERVENTIONS:
Procedure: Multidisciplinary tele-health intervention (physical therapy, neurologist, nurse, psychologist) — Non-pharmacological and pharmacological treatment provided by telemedicine plus in-office visits
  Other Names: Education
  Arms: Study group
Other: Standard in-office medical care — Non-pharmacological and pharmacological treatment provided in-office visits
  Arms: Control group

SUMMARY:
Falls in Parkinson's Disease (PD) are very frequent with often devastating consequences, increasing comorbidity, mortality, decreased quality of life and increased socio-health costs. In this national, single-center, single-blind, randomized, case-control study, non-demented patients with idiopathic PD with high risk of falling will be included. The main objective of this study is to determine the cost-effectiveness of a home-based, multidisciplinary tele-health intervention to decrease the risk of falling.

DETAILED DESCRIPTION:
In this study, PD patients using multidisciplinary tele-health intervention (study group) will be compared to age, gender-matched PD patients receiving the best standard in-office clinical management (control group). Both groups will be followed for 8 months.

The main outcome will be the comparison of incidence of falls between the study and control groups. Secondary outcomes will include the analysis of cost-effectiveness of multidisciplinary tele-health interventions.

The results of this study will allow us to study the feasibility of remote health care to prevent falls in patients with PD, allowing equity in the distribution and access to specialized health care.

ELIGIBILITY:
Inclusion Criteria:

* Non-demented patients
* Patients diagnosed with idiopathic Parkinson´s disease
* Patients able to walk with a Hoehn Yahr stage < 3

Exclusion Criteria:

* Non-ambulatory patients with Parkinson´s disease
* Patients diagnosed with significant comorbidity (psychiatric, systemic, hearing or visual disturbances) according to the investigator criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of falls reduction | 8 months
  Comparison of incidence of falls between the study and control groups by using diaries and wearable sensors
Feasibility | 8 months
  Number of virtual videoconferences completed

SECONDARY OUTCOMES:
Cost-effectiveness | 8 months
  To compare the medical and non-medical direct costs between the study and control groups by using structured questionnaires
Healt-related quality of life | 8 months
  To compare the PDQ-39 scores between the study and control groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No
MAIN RESULTS

REFERENCES:
- [Derived] Cubo E, Garcia-Bustillo A, Arnaiz-Gonzalez A, Ramirez-Sanz JM, Garrido-Labrador JL, Valinas F, Allende M, Gonzalez-Bernal JJ, Gonzalez-Santos J, Diez-Pastor JF, Jahouh M, Arribas J, Trejo J. Adopting a multidisciplinary telemedicine intervention for fall prevention in Parkinson's disease. Protocol for a longitudinal, randomized clinical trial. PLoS One. 2021 Dec 21;16(12):e0260889. doi: 10.1371/journal.pone.0260889. eCollection 2021. PMID 34932580